CLINICAL TRIAL: NCT03197038
Title: Exercise Training and Cognitive Function in Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ulf G. Bronas, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1217; P30AG022849 (NIH)
Record Dates: First submitted 2017-06-08; First posted 2017-06-23 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Cognitive Function, Preclinical; Chronic Kidney Diseases; Older Adults
Keywords: Cognitive function; Kidney Disease; Exercise; Older adults
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized, controlled design with a 1:1 allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based walking exercise (Experimental): Home-based exercise program: The exercise training group will participate in an educational session on exercise for CKD. Participants will receive a packet of information with an exercise prescription and a heart rate monitor that monitors the exercise. Participants will be asked to exercise (a brisk walk) at home, 3 times per week, for 30-60 minutes for 24 weeks. Participants will be contacted via phone biweekly or more frequently if they are behind the exercise routine, and the investigators will meet with them monthly to provide encouragement and progression of exercise, and to download the heart rate monitor.
  Interventions: Behavioral: Partially supervised home-based walking exercise
- Control (Active Comparator): The control group will receive standard instructions on exercise for patients with kidney disease similar to what is commonly done in clinical practice. The control group will not receive an exercise prescription or heart rate monitor. Participants will be contacted via phone biweekly to answer any questions and ensure continued study participation. The control group will not meet with the investigators monthly.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Partially supervised home-based walking exercise — Participants will be asked to exercise at home by walking at a moderate intensity. Each participant will receive an exercise prescription. Participants will receive a heart rate monitor. The heart rate monitors will be used to achieve a desired exercise intensity and to monitor adherence levels. The participants will receive biweekly to weekly phone calls, and monthly in person meetings will be used to address any barriers, provide encouragement, and progress the exercise.
  Arms: Home-based walking exercise
Behavioral: Control — Participants will be asked to exercise at home by walking at a moderate intensity. The participants will receive biweekly phone calls, but will not receive a heart rate monitor, individual exercise prescription, or meet with the investigators monthly.
  Arms: Control

SUMMARY:
Chronic kidney disease (CKD), affects over 45% of all individuals over 70 years of age. Patients with moderate CKD have more than a two-fold increased risk of cognitive impairment than those without CKD; furthermore, as many as 20-70% of patients with CKD have established cognitive impairment and overt dementia. The burden of cognitive impairment and dementia leads to functional decline and accelerated loss of independence, contributing to the tremendous individual, societal, and economic burden of CKD (i.e., 20% of Medicare expenditures in adults >65 years of age). There is no recommended treatment to prevent cognitive decline in CKD patients, and the few medications available for cognitive impairment have only short term modest effects. There is a critical need to evaluate therapies to forestall cognitive impairment, and maintain or improve cognitive functioning in older patients with CKD. To address this need, this study will test the hypothesis that older patients with moderate/severe CKD and pre-clinical cognitive impairment randomized to a 6-month home-based exercise program will improve cognitive function and MRI measured brain structure, compared to a usual care control group. This study will combine an assessment of cognition with MR imaging techniques to fully evaluate brain structure, blood flow, and behavior relationships at a level previously not conducted in this population

ELIGIBILITY:
Inclusion Criteria:

* English speaking men and women
* diagnosed stage 3-5 CKD (eGFR<60 to 15 ml/min);
* 60-80 years of age,
* self-experienced persistent decline in cognitive capacity determined as self-reported cognitive complaint (i.e., answering "yes" to the question: "Do you feel like your memory or thinking skills have gotten worse recently?" (before any clinical impairment of cognition has occurred)
* ability to undergo an MRI;
* no history of major head trauma.

Exclusion Criteria:

* • current/past diagnosis of neurological/psychiatric disorders;

  * any medications to improve cognition or mood;
  * Diagnosed Dementia or a score of <2 on the mini-cog assessment
  * Ischemic ulcerations or gangrene on the feet or legs;
  * Participating in a supervised exercise program with intent to increase fitness levels 3 days/week,
  * Requires assistive ambulation;
  * Limited exercise capacity due to conditions other than claudication

    * unstable angina,
    * Claudication
    * severe arthritis,
    * extreme dyspnea on exertion,
    * unstable coronary artery disease;
    * Class III-IV heart failure;
    * Current uncontrolled sustained arrhythmias,
    * severe/symptomatic aortic or mitral stenosis,
    * hypertrophic obstructive cardiomyopathy,
    * severe pulmonary hypertension,
    * active myocarditis/pericarditis,
    * thrombophlebitis,
    * recent systemic/pulmonary embolus (within 3 months);
  * Resting systolic BP >200 mmHg or resting diastolic BP >110 mmHg;
  * Revascularization procedures within the previous 6 months;
  * Any unforeseen illness or disability that would preclude exercise testing or training based on patient provider opinion;
  * Pregnancy
  * No diagnosis of CKD
  * One or more contraindication for MRI

    * cardiac pacemaker,
    * aneurysm clip,
    * cochlear implants,
    * shrapnel,
    * history of metal fragments in eyes,
    * neurostimulators,
    * diagnosed claustrophobia.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulf G Bronas, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bronas UG, Hannan M, Lash JP, Ajilore O, Zhou XJ, Lamar M. Exercise Training and Cognitive Function in Kidney Disease: Protocol for a Pilot Randomized Controlled Trial. Nurs Res. 2022 Jan-Feb 01;71(1):75-82. doi: 10.1097/NNR.0000000000000554. PMID 34570042

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Home-based Walking Exercise | Control
Started | 22 | 17
Completed | 18 | 17
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home-based Walking Exercise | Control | Total
Number analyzed (Participants) | 22 | 17 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 5 | 16
  >=65 years | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.68 (4.4) | 68.76 (5.7) | 67.6 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 19 | 14 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 14 | 28
  White | 7 | 3 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 17 | 39

OUTCOME MEASURES:

1. Primary Outcome: Composite Global Cognitive Function
Description: Determine the effect of a 6-month home-based exercise program on composite global cognitive functioning as determined by principal component analysis of immediate free recall of trials 1-5 on California verbal learning II, long-delay free recall and recognition, and memory discriminability, trail making test part A and part B, digit symbol substitution test, semantic and phonemic fluency, and Digit span subtest in older patients with kidney disease and preclinical cognitive impairment. A composite global cognitive score was created by converting the individual cognitive scores to standardized z scores and then averaging the standardized z scores. An increase in change from baseline to 6 months is considered an improvement.
Time Frame: Change from baseline in composite global cognitive function at 6 months
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 18 | 17
Z-score | .15 (.37) | .02 (.33)

2. Primary Outcome: Composite Executive Function
Description: A composite executive functioning score was created by converting 4 individual executive cognitive scores (verbal fluency FAS and animal summary score, digit span backward subtest, and TMT-B) to standardized z scores and then averaging the standardized z scores. A larger change in Z score is considered an improvement.
Time Frame: Change from baseline in composite executive function at 6 months
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 18 | 17
Z score | 0.21 (.47) | -.01 (.47)

3. Secondary Outcome: White Matter Integrity
Description: Whole brain white matter integrity was created by averaging the fractional anisotropy of 80 tracts using region of interest analysis. An increased change from baseline to 6 months in fractional anisotropy (a measure of directionality, 0 = no principle direction, 1 = one principle direction) is considered an improvement.
Time Frame: Change from baseline white matter integrity fractional anisotropy at 6 months
Population: Of the total sample of 39 participants, 31 participants were able to undergo MRI scans. Of these, four participants did not complete the study. Good quality data, without motion distortion , were available in 25 participants (two participants were excluded due to motion distortion) at baseline and follow-up and were included in the analysis (11 intervention participants and 14 control participants).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 11 | 14
units on a scale | -.002 (.02) | .003 (.01)

4. Secondary Outcome: Hippocampal Volume - Right
Description: Determine the effect of a 6-month exercise program on hippocampal volume. An increased change from baseline to 6 months in right hippocampal volume in cubic millimeters is considered an improvement.
Time Frame: Change from baseline hippocampal volume at 6 months.
Population: Of the total sample of 39 participants, 31 participants were able to undergo MRI scans. Of these, four participants did not complete the study. Good quality data, without motion distortion, were available in 21 participants (four participants were excluded due to motion distortion) at baseline and follow-up and were included in the analysis (9 intervention participants and 12 control participants).
Measure: Mean (Standard Deviation); unit: Cubic millimeters
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 9 | 12
Cubic millimeters | .003 (.0002) | .003 (.003)

5. Secondary Outcome: Cerebral Blood Flow
Description: Determine the effect of a 6-month exercise program on cerebral blood flow. Change in global cerebral blood measured in mL/100g/min from baseline to 6 months. An larger change is considered an improvement.
Time Frame: Change from baseline in cerebral blood flow at 6 months.
Population: Of the total sample of 39 participants, 31 participants were able to undergo MRI scans. Of these, four participants did not complete the study. Good quality data, without motion distortion, were available in 25 participants (two participants were excluded due to motion distortion) at baseline and follow-up and were included in the analysis (11 intervention participants and 14 control participants).
Measure: Mean (Standard Deviation); unit: mL/100gm/min
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 11 | 14
mL/100gm/min | 1.6 (9.8) | 0.3 (12.2)

6. Secondary Outcome: Vascular Health - Young's Elastic Modulus
Description: Vascular health was assessed by Young's Elastic Modulus (YEM) at the carotid artery. A larger negative change in YEM (measured in kilo pascal, stiffer artery=higher number) from baseline to 6 months is considered an improvement.
Time Frame: Change from baseline in vascular health indices at 6 months
Population: Of the total sample of 39 participants, four participants did not complete the study. Good quality data, without motion distortion, were available in 33 participants (two participants were excluded due to motion distortion) at baseline and follow-up and were included in the analysis (17 intervention participants and 16 control participants).
Measure: Mean (Standard Deviation); unit: Kilo pascals
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 17 | 16
Kilo pascals | -3,175 (9,428) | 1,279 (8,654)

7. Secondary Outcome: Cognitive Function - Total Cognition
Description: Determine the effect of a 6-month exercise program on cognitive function via the NIH toolbox
  This composite includes: Flanker, Dimensional Change Card Sort, Picture Sequence Memory, List Sorting and Pattern Comparison. This composite score is derived by averaging the standard scores of each of the measures, and then deriving standard scores based on this new distribution. An Age-Corrected Standard Score was used.
  Scale runs 140 to 23, a higher score means a better outcome. An increased change from baseline to 6 months is considered an improvement
Time Frame: Mean change from baseline to 6 months.
Population: Data was collected in a sub-sample (n=12) to provide pilot data on the NIH-toolbox as part of an administrative supplement. Of the 12 participants that were part of the sub-sample, two did not complete the study. Baseline and follow-up data was available in 10 participants (6=intervention, 4=control).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 6 | 4
Score on a scale | 8 (7.4) | 11 (7.6)

8. Secondary Outcome: Motor Function - Grip Strength
Description: Determine the effect of a 6-month exercise program on motor function via the NIH toolbox. Age corrected grip strength on a standard scale. Standard scale 140-23, higher score is better. An increased change from baseline to 6 months is considered an improvement.
Time Frame: Change from baseline in NIH toolbox motor function indices at 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 6 | 4
Score on a scale | 3 (6.2) | -2.5 (7.2)

9. Secondary Outcome: Vascular Health - Pulse Wave Velocity
Description: Vascular function indices of vascular health was assessed using pulse wave velocity of the aorta in meters/second (higher number =more stiff aorta). A larger negative change from baseline to 6 months is considered an improvement.
Time Frame: 6 Months
Population: Of the 39 participants that were enrolled, four did not complete the study. Good quality data without motion distortion at baseline and follow up was available in 30 participants (15=intervention, 15=control).
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 15 | 15
Meters per second | -.01 (1.1) | .21 (.92)

10. Secondary Outcome: Vascular Health - Augmentation Index
Description: Vascular function indices of vascular health was assessed using augmentation index at the carotid artery (in percentage, higher percent=more stiff artery). A larger negative change from baseline to 6 months is considered an improvement.
Time Frame: 6 Months
Population: Of the 39 participants enrolled, four did not complete the study. Good quality data without motion distortion at baseline and follow-up was available in 34 participants (18=intervention, 16=control).
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 18 | 16
Percentage | -2.6 (12.1) | 3.3 (16.6)

11. Secondary Outcome: Cognitive Function - Fluid Cognition
Description: Determine the effect of a 6-month exercise program on cognitive function via the NIH toolbox. Fluid cognition.
  This composite includes: Flanker, Dimensional Change Card Sort, Picture Sequence Memory, List Sorting and Pattern Comparison. This composite score is derived by averaging the standard scores of each of the measures, and then deriving standard scores based on this new distribution. An Age-Corrected Standard Score was used. A larger change from baseline to 6 months is considered an improvement.
  Scale runs 140 to 23, a higher score means a better outcome.
Time Frame: Mean change from baseline to 6 months.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 6 | 4
Score on a scale | 5.2 (12.2) | 11 (8.9)

12. Secondary Outcome: Cognitive Function - Crystalized Cognition
Description: Change from baseline in NIH toolbox cognitive function indices at 6 months. Crystalized cognition.
  This composite includes : Flanker, Dimensional Change Card Sort, Picture Sequence Memory, List Sorting and Pattern Comparison. This composite score is derived by averaging the standard scores of each of the measures, and then deriving standard scores based on this new distribution. An Age-Corrected Standard Score was used.
  An larger change from baseline to 6 months is considered an improvement. Scale runs 140 to 23, a higher score means a better outcome.
Time Frame: Mean change from baseline to 6 months.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 6 | 4
Score on a scale | 7.7 (7.5) | 8.3 (7.1)

13. Secondary Outcome: Motor Function - Balance
Description: Determine the effect of a 6-month exercise program on motor function via the NIH toolbox. Change in balance age corrected standard score from baseline to 6-months (23-140, higher score is better). A larger change is considered an improvement.
Time Frame: 6 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 6 | 4
Score on a scale | -6 (8.5) | -8 (25)

14. Secondary Outcome: Motor Function - Dexterity
Description: Determine the effect of a 6-month exercise program on motor function via the NIH toolbox. Hand dexterity was determine using age corrected standard scale in the dominant hand. A larger change from baseline to 6 months is considered an improvement.
  Standard scale range 140-23, higher score is better.
Time Frame: 6 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 6 | 4
Score on a scale | 1.2 (4.5) | 1.8 (15.5)

15. Secondary Outcome: Resting Global Connectivity
Description: Resting global connectivity measured and averaged across 132 regions. A larger change from baseline to 6 months is considered an improvement. Connectivity is a correlation (increased connectivity=higher correlation)
Time Frame: Change from baseline at 6 months
Population: Resting global connectivity was collected in a sub-sample (n=12) to provide pilot data. Of the 12 participants that were part of the sub-sample, two did not complete the study. Good quality data without motion distortion at baseline and follow-up was available in 10 participants (5=intervention, 5=control).
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 5 | 5
Z-score | .0047 (.0356) | -.0310 (.019)

16. Secondary Outcome: Hippocampal Volume - Left
Description: Determine the effect of a 6-month exercise program on hippocampal volume. An larger change from baseline to 6 months in left hippocampal volume (cubic millimeters) is considered an improvement.
Time Frame: Change from baseline at 6 Months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Cubic millimeters
Arm/Group | Home-based Walking Exercise | Control
Number analyzed (Participants) | 9 | 12
Cubic millimeters | -.0001 (.0002) | .0 (.0001)

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Home-based Walking Exercise | Control
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/17
Other Adverse Events (participants affected / at risk) | 14/22 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home-based Walking Exercise (N=22) | Control (N=17)
Transient ischemic attack (Vascular disorders) | 1 (1) | 0 (0) — An intervention participant was diagnosed with a transient ischemic attack (TIA). It was determined that this event was unrelated to study procedures and that no protocol revisions were required. The participant was discontinued from the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home-based Walking Exercise (N=22) | Control (N=17)
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
ED visit: non-serious illness (General disorders) | 3 (3) | 4 (4)
ED visit: non-specific chest pain (Cardiac disorders) | 1 (1) | 4 (4)
ED visit - fall with head injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Participant fell out of bed at home. Unrelated to study participation.
ED visit - blood pressure (Cardiac disorders) | 1 (1) | 0 (0)
Dental surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Home repair accident (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Drywall well on participant.
Urgent care visit: Calf pain, possible DVT (Vascular disorders) | 1 (1) | 0 (0)
ED visit: feeling of weakness (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Possible anemia
Prostate and hernia surgery (Surgical and medical procedures) | 2 (2) | 1 (1)
Low ejection fraction (Cardiac disorders) | 1 (1) | 0 (0)
Calf muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT03197038/Prot_SAP_000.pdf